CLINICAL TRIAL: NCT03025672
Title: Evaluation of the Cost of a Nosocomial Infection With Clostridium Difficile
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: OBS-021
Record Dates: First submitted 2017-01-10; First posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Cross Infection; Clostridium Difficile Infection
MeSH Terms: conditions — Cross Infection; Clostridium Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- clostridium difficile: Patients that have been infected by clostridium difficile during their stay in hospital
- no clostridium difficile: Patients that have not been infected during their stay in hospital.

SUMMARY:
Clostridium difficile is the first cause of nosocomial infectious diarrhea, due to its mode of transmission and its resistance in the environment.

Nosocomiality is defined by the apparition of an infection 48 hours after the patient's hospitalization. Clostridium difficile contamination occurs oro-fecally and is transmitted directly through the hand or from the contaminated environment (during care or not). By implementing prevention and optimal treatment, nosocomial infections are preventable.

A clostridium difficile infection causes an additional cost of patient care for the hospital. This additional cost is principally due to the increase of the length of the stay. It varies according to patient risk factors,and also according to the reason of the hospitalization and can vary from 300 euros (~317$) to more than 25.000 euros (26.460$).

By determining the increase in the length of the stay and the additional cost due to a clostridium difficile infection in the GHICL (Groupement des Hôpitaux de l'Institut Catholique de Lille), prevention will be valued and measures against those infections should be easier to set up.

The main objective of this study is to evaluate the additional cost of an infection by clostridium difficile.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have stayed in an hospital of the GHICL between January 2013 and September 2015.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that have stayed in an hospital of the GHICL in 2013 and 2014
Sampling Method: Non-Probability Sample
Enrollment: 10445 (Actual)
Dates: Start 2015-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Difference between patient cost and income for the hospital based on the PMSI rate. | Day 1
  The difference between the real cost of the patient stay, included the additional costs due to clostridium difficile infection, and the public funding (calculated using the PMSI) for this stay will be computed.

IPD SHARING:
Plan to Share IPD: No